CLINICAL TRIAL: NCT03974113
Title: ATLAS-PEDS: An Open-label, Multinational Study of Fitusiran Prophylaxis in Male Pediatric Subjects Aged 1 to Less Than 12 Years With Hemophilia A or B
Brief Title: Fitusiran Prophylaxis in Male Pediatric Subjects Aged 1 to Less Than 12 Years With Hemophilia A or B
Acronym: ATLAS-PEDS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFC15467; U1111-1223-4368 (Registry Identifier: ICTRP); 2024-512501-76 (Registry Identifier: CTIS); 2019-000679-18 (EudraCT Number)
Record Dates: First submitted 2019-06-03; First posted 2019-06-04 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — fitusiran

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fitusiran (Experimental): Participants will receive a selected dose of fitusiran at regular intervals, as per study protocol
  Interventions: Drug: Fitusiran

INTERVENTIONS:
Drug: Fitusiran — Pharmaceutical form:Solution for injection-Route of administration:Subcutaneous
  Other Names: SAR439774

SUMMARY:
Primary Objective:

- To confirm appropriate dose levels of fitusiran when administered to male pediatric participants (ages 1 to <12 years of age) with severe hemophilia A or B

Secondary Objectives:

* To characterize the safety and tolerability
* To determine fitusiran plasma concentrations at selected time points

DETAILED DESCRIPTION:
The estimated total time on study is up to 256 weeks for participants who roll over into the extension study and up to 280 weeks for participants who do not roll over into the extension study (due to the requirement for up to an additional 6 months of follow-up for monitoring of AT levels).

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 1 to <12 years at the time of enrollment.
* Severe hemophilia A or B (Factor VIII (FVIII) <1% or Factor IX (FIX) ≤2%)
* Participants must have inhibitory antibodies to FVIII or FIX and must meet one of the following Nijmegen-modified Bethesda assay results criteria:

  * Inhibitor titer of ≥0.6 BU/mL at screening, OR
  * Inhibitor titer of <0.6 BU/mL at screening with medical record evidence of 2 consecutive titers ≥0.6 BU/mL, OR
  * Inhibitor titer of <0.6 BU/mL at screening with medical record evidence of 1 inhibitor titer ≥0.6 BU/mL and a history of anamnestic response or severe allergic reaction (anaphylaxis or nephrotic syndrome)
* Adequate peripheral venous access, as determined by the Investigator, to allow the blood draws required by the study protocol
* Weight requirements at the time of enrollment: 8 to <45 kg
* Willing and able to comply with the study requirements and to provide signed written informed consent obtained from parent(s)/legal guardian (hereinafter the "parent") and written or oral assent obtained from participant, per local and national requirements

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Known co-existing bleeding disorders other than hemophilia A or B
* Antithrombin (AT) activity <60% at Screening
* Co-existing thrombophilic disorder
* Clinically significant liver disease
* Active Hepatitis C virus infection
* Acute or chronic Hepatitis B virus infection
* Acute Hepatitis A or hepatitis E infection
* HIV positive with a CD4 count of <400 cells/μL
* History of arterial or venous thromboembolism, unrelated to an indwelling venous access
* Inadequate renal function
* History of multiple drug allergies or history of allergic reaction to an oligonucleotide or N-Acetylgalactosamine (GalNAc)
* Subjects with central or peripheral indwelling catheters, with history of venous access complications leading to hospitalization and/or systemic anticoagulation therapy.
* History of intolerance to subcutaneous (SC) injection(s)
* Use of emicizumab (Hemlibra®) within 6 months prior to screening
* Any other conditions or comorbidities that would make the patient unsuitable for enrollment or could interfere with participation in or completion of the study, per Investigator judgment

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 1 Year to 11 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Plasma antithrombin (AT) activity levels | Day 1 to the AT analysis time point at the optimal therapeutic dose (approximately 256 weeks)
  Characterize the AT activity at the optimal therapeutic dose

SECONDARY OUTCOMES:
Number of participants reported with adverse events | Up to 280 weeks (up to 256 weeks of treatment + up to 24 weeks of AT follow up)
  Number of participants reported with treatment-emergent adverse events (TEAEs)
Fitusiran plasma concentrations | Day 1 and Day 85
  Plasma samples will be collected for measurement of plasma concentrations of fitusiran at specific time points post dose on Day 1 and pre dose on Day 85

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (16):
- United States (4):
  - Children's Hospital Los Angeles Site Number : 8400002, Los Angeles, California
  - Hackensack University Medical Center- Site Number : 8400008, Hackensack, New Jersey
  - University Hospitals of Cleveland- Site Number : 8400007, Cleveland, Ohio
  - Penn State Milton S. Hershey Medical Center- Site Number : 8400006, Hershey, Pennsylvania
- Canada (2):
  - Investigational Site Number : 1240001, Hamilton, Ontario
  - Investigational Site Number : 1240002, Ottawa, Ontario
- India (4):
  - Investigational Site Number : 3560006, Bangalore
  - Investigational Site Number : 3560002, Mumbai
  - Investigational Site Number : 3560001, Pune-411011
  - Investigational Site Number : 3560004, Vellore
- Italy (2):
  - Investigational Site Number : 3800002, Florence
  - Investigational Site Number : 3800001, Milan
- Investigational Site Number : 7240002, Madrid, Madrid, Comunidad de, Spain
- Turkey (Türkiye) (3):
  - Investigational Site Number : 7920001, Adana
  - Investigational Site Number : 7920002, Istanbul
  - Investigational Site Number : 7920003, Izmir

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org